CLINICAL TRIAL: NCT01190683
Title: Skeletal Muscle Strength,Bone Mineral Homeostasis and Th1 and Th2 Cytokines Expression in Asian Indians With Chronic Hypovitaminosis D Before and After Oral Cholecalciferol Supplementation
Brief Title: Vitamin D and Muscle Strength and Surface (Electromyography) EMG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indian Council of Medical Research (Other Government)
Responsible Party: Dr Ravinder Goswami, Additional Professor, Department of Endcrinology and Metabolism, All India Institute of Medical Sciences, New Delhi 110029
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: IEC/NP-216/2010
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2010-08

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D; Calcium Carbonate; Calcium; Lactose; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- cholecalciferol (Active Comparator): cholecalciferol 60,000IU/week for first eight weeks followed by 60,000 IU every 15 days for four months along with calcium placebo
  Interventions: Drug: Cholecalciferol; Drug: Calcium Carbonate; Drug: cholecalciferol and calcium carbonate; Other: lactose granules and tablets
- Calcium carbonate (Active Comparator): two tablets of calcium carbonate daily equivalent to 1 gm of elemental calcium for six months along with vitamin D placebo
  Interventions: Drug: Calcium Carbonate; Drug: cholecalciferol and calcium carbonate; Other: lactose granules and tablets
- oral calcium and cholecalciferol (Active Comparator): 60,000 IU of cholecalciferol every week for ist eight week and then 60,000IU every 15 days for next four months along with 1 gm of elemental calcium ever day for six months
  Interventions: Drug: cholecalciferol and calcium carbonate; Other: lactose granules and tablets
- lactose (Placebo Comparator): identical placebos
  Interventions: Other: lactose placebo; Other: lactose granules and tablets

INTERVENTIONS:
Drug: Cholecalciferol — 60,000 IU/week for ist eight weeks followed by 60,000 IU every 15 days for four months
  Other Names: Vitamin D
  Arms: cholecalciferol
Drug: Calcium Carbonate — two tablets of calcium carbonate daily containing 1 gm of elemental calcium for six months
  Other Names: Calcium
  Arms: Calcium carbonate; cholecalciferol
Drug: cholecalciferol and calcium carbonate — 60,000 IU of cholecalciferol for first eight weeks and then 60,000IU for next four months along with 1 gm of elemental calcium daily for six months
  Other Names: vitamin D and calcium carbonate
  Arms: Calcium carbonate; cholecalciferol; oral calcium and cholecalciferol
Other: lactose placebo — similar number of granules and tablets as active group
  Other Names: lactose
  Arms: lactose
Other: lactose granules and tablets — one sachet every week for eight weeks followed by two sachets every month along with two lactose tablets daily

SUMMARY:
Vitamin D deficiency is widely prevalent in India. Serum 25(OH)D levels are <20 ng /ml in up to 90% of them. Recently, in a randomized control trial, investigators have shown that dual cholecalciferol and calcium supplementation lead to significant improvement in hand grip strength and distance covered during six minutes walk test. Present study is being taken to further understand the functional significance of 25(OH)D in terms of its effect on Skeletal muscle strength including surface electromyography (EMG) in a larger cohort involving approximately 200 subjects. The impact of calcium and vitamin D supplementation would be assessed by supplementing them alone and in combination. Besides, the investigators would also assess impact of above supplementation on Th1/Th2 cytokines expression in the peripheral mononuclear cells.

DETAILED DESCRIPTION:
Vitamin D is an essential nutrient that plays an important role in calcium metabolism and bone health. In recent years, biomarkers like PTH, calcium absorption have been used to define relevant biological indices of vitamin D nutritional status. Several studies from India have shown wide prevalence of vitamin D deficiency (VDD) in India. Goswami et al studied serum 25 (OH)D levels and its functional significance in apparently healthy subjects residing in Delhi and showed low serum 25(OH)D values in all the groups (Am J Clin Nutr 2000). Its functional significance is currently under evaluation.

Relevant studies assessing functional significance of VDD in Asian Indians are summarized below (Am J Clin Nutr 2000).

A) Goswami et al while reporting low serum 25(OH) D concentrations in healthy subjects in Delhi, showed a higher serum PTH levels & significant inverse relation between serum 25(OH) D and PTH levels ( r = -0.6303, p < 0.001) in all the three groups (soldiers, physicians & nurses, depigmented persons) studied in winter (Am J Clin Nutr 2006) B) Effects on BMD Recently,we have analyzed relationship between BMD and serum 25(OH) D in 105 apparently healthy Asian Indian. The cohort of 105 subjects was split into 2 groups at a serum 25(OH) D cutoff of 9.0 ng/mL. The mean serum iPTH was significantly higher in the group 1 (<9.0 ng/ml)than in the group 2 subjects (53.1±31.3 and 39.3±17.5 pg/mL, respectively; P=0.012).The mean BMD values of the total hip, including femoral neck, trochanter, and intertrochanter, were significantly (P = 0.001) lower in group 1 than in group 2.

C) Effect of VDD on intestinal calcium absorption in Asian Indians with chronic hypovitaminosis D and its change after cholecalciferol supplementation was studied recently at our Department of Endocrinology and Metabolism. Study subjects were 29 apparently healthy volunteers [17 M, 12 F, mean (SD) age = 28.4 ± 6.4 year] with low serum 25(OH)D levels [mean (SD) = 7.6 ± 4.8 ng/ml]. Intestinal calcium absorption was assessed by 'calcium load test' (PAK test) (10) using 1 gm of oral elemental calcium load before and after (n = 26) supplementation with oral cholecalciferol (60,000 IU/week for eight weeks). This study showed that the vitamin D Deficiency is physiologically relevant in terms of intestinal calcium absorption in Asian Indians (Journal of Human Nutrition and dietetics 2010).

Recently in a randomized control trial we have shown significant improvement in the muscle strength and walking distance after dual supplementation with cholecalciferol and calcium (Clin Endocrinol 2010). In the current study we plan to study this aspect further by recruiting four groups to study the effect of calcium and vitamin D supplementation alone or in combination as a dual supplementation. Baseline evaluation (Before vitamin D supplementation) would include serum total calcium, inorganic phosphorus, alkaline phosphatase, intact PTH and 25(OH) D assays, hand grip muscle strength and surface EMG testing. Hand grip would be done will be done using a computerized dynamometer in the Department of Physical Medicine and Rehabilitation under the guidance of Professor U Singh, Head, Department of Physical Medicine & Rehabilitation, AIIMS. Handgrip strength will be measured in right hand by dynamometer. The average of two measurement of grip strength will be used for analysis (in kg).

The physical performance will be tested by performing 6 - minute walk test using standard protocol and results will be interpreted in terms of 6 minute walk distance in meters and degree of shortness of breath using modified Borg dyspnea scale.

The mRNA expression Th1 and Th2 cytokines would be assessed in the PBMC drawn from 5 ml of the peripheral blood using the real time PCR.

Vitamin D supplementation

All the subjects will be randomized into three treatment groups and one placebo group in a double blind manner. Random code would be generated by a investigator, who will not be involved in distribution of medicines and assessment of the muscle strength Active drug would be calcium (two tablets of calcium carbonate each containing 500 mg of elemental calcium/day, and 60,000 IU of cholecalciferol/week obtained from the commercial source. The inactive drug would be lactose containing identical placebo obtained from the same source. All study subjects will be provided with packets containing four sachets of cholecalciferol (each containing 60000 IU vitamin D3; Cadila Pharmaceutical, India) /placebo; and sixty tablets of calcium carbonate (500mg elemental calcium & 250 IU vitamin D3; Elder Pharmaceutical, India)/placebo. First dose will be supervised. Subjects will be counseled for daily intake of two tablets of calcium carbonate and weekly intake of a cholecalciferol sachet and follow up at completion of 4 weeks. Similar packets will be given after 4 weeks of follow up. Drug compliance will be assessed by counting the empty sachets. After eight week subjects will be provided daily two tablets of calcium carbonate containing 500 mg elemental calcium each and two sachets of cholecalciferol every month for four months.

Assessment at 8 weeks and 6 months would include serum intact PTH & 25(OH) D levels estimation, skeletal muscle strength testing, and 6 minute walk test and Th1/Th2 analysis

Safety of Proposed Interventions Cholecalciferol dose of 60000 IU/week × 8 weeks has been considered safe to be used in healthy subjects, as shown in our recent studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Residence of Delhi
* Commitment for follow-up at 8 weeks, 6 months.
* Consent for supplementation

Exclusion Criteria:

* Subjects taking drugs, which can affect bone mineral metabolism such as glucocorticoids, antitubercular, antiepileptics, levothyroxine, bisphosphonates
* Chronic renal or liver disorder
* Chronic diarrhea

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Improvement in Muscle strength | six months
  To assess change in upper and lower limb muscle strength by measiung hand grip, walking distance during six months of supplemnation with oral calcium carbonate alone, oral cholecalciferol alone, and dual supplemenation with oral cholecalciferol and calcium carbonate

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ravinder Goswami, MD, DM, Principal Investigator — Associate Professor, Department of Endcorinology and Metabolism, All India Institute of Medical Sciences, New Delhi 110029, India; Dr U Singh, MBBS, MD, Principal Investigator — Professor and Head, Department of Physcical Medicine and Rehablitation, All India Institute of Medical Sciences, New Delhi 110029, India; Dr Nandita Dupta, PhD, Principal Investigator — Additional Professor, Department of Endocrinology and Metabolism, All India Institute of Medical Sciences, New delhi 110029, India; Dr Manjari Tripathy, DM, Principal Investigator — Associate Professor, Department of Neurology, All India Institute of Medical Sciences, New Delhi 110029, India; Dr Manju Vatsa, Principal Investigator — Principal, College of Nursing, All India Institute of Medical Sciences, New Delhi 110029, India